CLINICAL TRIAL: NCT00678197
Title: Philippine Child Health and Policy Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: John W. Peabody, University of California San Francisco
Purpose: Health Services Research
Other Study IDs: R01HD042117 (NIH); R01HD042117 (NIH)
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Childhood Illness
Keywords: Quality of care; Access to care; Health Outcomes

ARMS (3):
- A (Experimental)
  Interventions: Other: Access Intervention
- B (Experimental)
  Interventions: Other: Bonus/Pay-for-Performance Intervention
- C (No Intervention)

INTERVENTIONS:
Other: Access Intervention
  Arms: A
Other: Bonus/Pay-for-Performance Intervention
  Arms: B

SUMMARY:
The long-term consequences of poverty on child health, including cognitive development, are one of the world's great tragedies. In the Philippines, diarrhea, acute lower respiratory infections, and the attendant problems of malnutrition, are the leading causes of childhood illness. The Philippine government plans to launch a broad national Health Sector Reform Agenda (HSRA) that will address the problems of poverty and illness in children. The introduction of these reforms provides an exceptional opportunity to conduct a social experiment. Four institutions, already involved in the design and implementation of the HSRA, plus leading experts in international health, government, and health measurement will collaborate on this project to collect longitudinal data and measure the impact of HSRA reforms on child health outcomes in a population. We will measure the health impacts of two experimental interventions: (1) expansion of health insurance coverage, and (2) capitation of providers. Our research will measure the impact of health reforms on the physical and cognitive health outcomes of children age 0-4. We will use a block design of 21 sites throughout the Philippines: seven for each of the two interventions, and seven matched controls. We will measure the quality of clinical practice using vignettes and will measure health outcomes using objective clinical tests. We will also use an advanced sampling strategy and panel data to link clinical practice with population health outcomes. This unparalleled research opportunity will yield significant insights about specific, unanswered questions of tremendous importance: Does health care serve as a social intervention that ameliorates the effects of morbidity and malnutrition on cognitive development? How effective are government policies at creating incentives to improve the quality of clinical practice? Do financial and organizational policies actually lead to better health and developmental outcomes? The results from this study will provide insights into the linkages between increased access, high quality care, and health outcomes in children.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting to participating hospitals

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2003-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09

CONTACTS AND LOCATIONS:
Locations (1):
- Manila, Philippines

REFERENCES:
- [Derived] Peabody JW, Florentino J, Shimkhada R, Solon O, Quimbo S. Quality variation and its impact on costs and satisfaction: evidence from the QIDS study. Med Care. 2010 Jan;48(1):25-30. doi: 10.1097/MLR.0b013e3181bd47b2. PMID 20009777
- See also: Related Info — http://qids.ph